CLINICAL TRIAL: NCT05496426
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Trial Evaluating the Safety and Efficacy of KL130008 Capsule in Patients With Severe Alopecia Areata
Brief Title: A Study of KL130008 in Adults With Severe Alopecia Areata
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KL223-II-05; CTR20221881 (Registry Identifier: KL223-II-05)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Hypotrichosis; Hair Diseases
MeSH Terms: conditions — Alopecia Areata; Hypotrichosis; Hair Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KL130008 capsule High Dose (Experimental): KL130008 capsule administered orally
  Interventions: Drug: KL130008/Placebo
- KL130008 capsule Middle Dose (Experimental): KL130008 capsule administered orally
  Interventions: Drug: KL130008/Placebo
- KL130008 capsule Low Dose (Experimental): KL130008 capsule administered orally
  Interventions: Drug: KL130008/Placebo
- Placebo (Placebo Comparator): Placebo administered orally
  Interventions: Drug: KL130008/Placebo

INTERVENTIONS:
Drug: KL130008/Placebo — Drug: KL130008 Drug: Placebo

SUMMARY:
The purpose of this study is to assess KL130008 is safe and effective in adults with severe alopecia areata

DETAILED DESCRIPTION:
This is a multi-center Phase 2 study to evaluate the safety and effectiveness of an investigational drug in adults (≥18 years and ≤65 years) who have 50% or greater scalp hair loss, including alopecia totalis (AT) and alopecia universalis (AU).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with the age of ≥18 and ≤ 65 years old at the time of informed consent.
2. Able to understand the procedures and methods of this study, and will to provide a signed and dated informed consent form.
3. Diagnosed alopecia areata(AA) without other reasons caused alopecia.
4. Have severe AA, as determined by all of the following:Current AA episode of more than 6 months' duration and hair loss encompassing ≥50% of the scalp, including alopecia totalis (AT) and alopecia universalis (AU);No spontaneous improvement over the past 6 months;Current episode of severe AA of less than 8 years.
5. All women of childbearing potential and all men must be willing to use at least one highly effective method of contraception from the signing of informed consent, throughout the duration of the study, and for 3 months after the last dose of investigational drugs.

Exclusion Criteria:

1. Known history of anaphylaxis to any of the ingredients and/or other similar products.
2. Participated in a clinical trial of any drug or medical device and has used an investigational product (including placebo and control group) or treatment within 1 month or 5 half-lives before randomization.
3. Previously treated with JAK inhibitors.
4. Corticosteroids, finasteride, minoxidil,topical immunotherapy treated within 8 weeks before randomization.
5. Diphenylcyclopropenone (DPCP), HMGCoA reductase inhibitor, Chinese herbal medicine treated within 4 weeks before randomization.
6. With other diseases: acute "diffuse" type of AA, lymphoproliferative disease, tumor, severe chronic gastrointestinal disease, thyroid disorders, serious cardiovascular disease.
7. Subjects with evidence of clinical laboratory abnormalities at screening that, in the opinion of the investigator, may affect the safety of subjects or the interpretation of study results: Hemoglobin level < 10.0 g/dL. Absolute white blood cell (WBC) count /absolute neutrophil count (NEUT)/absolute lymphocyte count(LYMPH)<LLN. Aspartate aminotransferase (AST), or alanine aminotransferase (ALT) > 2 × ULN, total bilirubin(TBIL)>1.5 × ULN. QTcF> 450ms. Subjects with eGFR ≤ 60 mL/min based on Cockcroft-Gault calculation.
8. The subject had or currently has a severe infection, and had a severe infection judged by the investigator within 1 month before randomization: HBV, TP-Ab, HIV, HCV, TB positive.
9. Subjects who are unsuitable to the trial, as identified by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 20 [ Time Frame: Week 24 ] | Week 24
  Percentage of Participants Achieving SALT ≤ 20

SECONDARY OUTCOMES:
Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 20 [ Time Frame: Week 36 ] | Week 36
  Percentage of Participants Achieving SALT ≤ 20
Percent Change from Baseline in SALT score [ Time Frame: Baseline, Week 24, 36 ] | Week 24, 36
  Percent change from baseline in SALT score
Percentage of Participants Achieving 50% Improvement of Severity of Alopecia Tool (SALT50) [ Time Frame: Week 24, 36 ] | Week 24, 36
  Percentage of participants achieving SALT50
Percentage of Participants Achieving 75% Improvement of Severity of Alopecia Tool (SALT50) [ Time Frame: Week 24, 36 ] | Week 24, 36
  Percentage of participants achieving SALT75
Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 10 [ Time Frame: Week 24, 36 ] | Week 24, 36
  Percentage of Participants Achieving SALT ≤ 10
Measure for Eyebrow (EB) Hair Loss 0 or 1 with ≥2-point Improvement from Baseline [ Time Frame: Week 24, 36 ] | Week 24, 36
  EB hair loss 0 or 1 with ≥2-point Improvement from Baseline
Measure for Eyelash (EL) Hair Loss 0 or 1 with ≥2-point Improvement from Baseline | Week 24, 36
  EL hair loss 0 or 1 with ≥2-point Improvement from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xingqi Zhang, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No